CLINICAL TRIAL: NCT02186808
Title: Procera-Bridge Zirconia - A Clinical Study
Brief Title: T-116_Procera-Bridge Zirconia - A Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nobel Biocare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T-116
Record Dates: First submitted 2014-06-27; First posted 2014-07-10 (Estimated); Results first posted 2016-04-25 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-09

CONDITIONS: Partial Edentulism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Procera® Bridge Zirconia (Other): Patients planned for treatment with a tooth-supported 3 to 4-unit bridge in any position of the maxilla or the mandible.
  Interventions: Device: Procera® Bridge Zirconia

INTERVENTIONS:
Device: Procera® Bridge Zirconia — Patients planned for treatment with a tooth-supported 3 to 4-unit bridge in any position of the maxilla or the mandible.

SUMMARY:
The objective of the study is to evaluate the clinical performance of Procera® Bridge Zirconia veneered with NobelRondo Zirconia.

DETAILED DESCRIPTION:
The study was designed to be an open, 5-year, prospective, multi-center clinical post-market study. The objectives of this clinical study were that industrial centrally produced 3- or 4-unit bridges of yttrium-oxide partially-stabilized (Y-TZP) zirconia (Procera Zirconia) in combination with the veneering ceramic material NobelRondo will show sufficient CDA ratings (90% R+S) and a sufficient survival rate after 1 and 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for treatment with a tooth-supported 3 to 4-unit bridge in any position of the maxilla or the mandible
* Indication: same indication as for metal supported bridges
* Obtained informed consent from the patient

Exclusion criteria

* Currently known alcohol, drug or medication abuse, judged by the investigator, which might influence the follow-up program
* Patients where a bridge part connection area of 3 mm of diameter is not possible to obtain (short clinical crowns)
* Mobility of the abutment teeth exceeding grade I
* Patients with pathologic pocket formation at abutment teeth
* Patients with complete dentures in the opposing jaw
* Patients with a removable partial denture in the same jaw

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Association, C.D., Quality Evaluation for Dental Care. Guidelines for the Assessment of Clinical Quality and Professional Performance. Los Angeles: CDA, 1977.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Procera® Bridge Zirconia
Started | 80
Completed | 67
Not Completed | 13

BASELINE CHARACTERISTICS:
Arm/Group | Procera® Bridge Zirconia
Number analyzed (Participants) | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 71
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 32

OUTCOME MEASURES:

1. Primary Outcome: Success Rate of Bridge Procera Bridge Zirconia
Description: The CDA index (1) is Romeo or Sierra at delivery and remains so up to 1 year post loading.
Time Frame: prosthesis delivery, 1 year
Population: 78 patients were treated in total. 4 of the patients received two bridges (which is complaint with the protocol). Therefore there are more bridges than patients.
Measure: Number; unit: percentage of successful implants
Units Other Than Participants: bridges
Arm/Group | Procera® Bridge Zirconia
Number analyzed (Participants) | 78
Number analyzed (bridges) | 82
percentage of successful implants | 100
Statistical Analysis 1: Comparison: Procera® Bridge Zirconia; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Success Rate of Bridge Procera Bridge Zirconia
Description: The CDA index (1) is Romeo or Sierra at delivery and remains so 5 year post loading.
Time Frame: prosthesis delivery, 5 years
Population: 5 year data. Not all initially treated patients could be followed over the 5 years.
Measure: Number; unit: percentage of successful implants
Units Other Than Participants: Number of Bridges analyzed
Arm/Group | Procera® Bridge Zirconia
Number analyzed (Participants) | 67
Number analyzed (Number of Bridges analyzed) | 69
percentage of successful implants | 95.8

ADVERSE EVENTS:
Arm/Group | Procera® Bridge Zirconia
Serious Adverse Events (participants affected / at risk) | 3/80
Other Adverse Events (participants affected / at risk) | 38/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Procera® Bridge Zirconia (N=80)
Cardiac arrhytmia (Cardiac disorders) | 1 (1) — Deceased, no evidence for a device related complication is reported.
Heart disease (Cardiac disorders) | 1 (1) — Deceased, no evidence for a device related complication is reported.
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Deceased, no evidence for a device related complication is reported.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Procera® Bridge Zirconia (N=80)
Porcelain fractures (Surgical and medical procedures) | 22 (27)
occlusal adjustments (Surgical and medical procedures) | 14 (15)
Periodontal problems (Surgical and medical procedures) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No